CLINICAL TRIAL: NCT00640926
Title: A Phase 2, Multicenter, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of RX-1741 in the Treatment of Adult Patients With Mild to Moderate Severity of Community-Acquired Pneumonia (CAP)
Brief Title: Safety and Efficacy Study of Oxazolidinone to Treat Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RX-1741-201
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Community-Acquired Pneumonia (CAP)
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — radezolid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Radezolid 300 mg
  Interventions: Drug: Radezolid
- 2 (Experimental): Radezolid 450 mg
  Interventions: Drug: Radezolid
- 3 (Experimental): Radezolid 450 mg BID
  Interventions: Drug: Radezolid

INTERVENTIONS:
Drug: Radezolid — 300 mg/day, orally for 7-10 days
  Other Names: RX-1741
  Arms: 1
Drug: Radezolid — 450 mg/day orally for 7-10 days
  Other Names: RX-1741
  Arms: 2
Drug: Radezolid — 900 mg/day orally for 7-10 days
  Other Names: RX-1741
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether RX-1741, an oxazolidinone antibiotic, is safe and effective in the treatment of mild to moderate community acquired pneumonia (CAP).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with mild to moderate CAP.
* Adult men and women ≥18 years.
* Females must be post-menopausal for at least 1 year or surgically sterile (hysterectomy or tubal ligation).
* Sexually active males must use a barrier method of birth control during and for 30 days after the study. Their female partner should also use an additional reliable method of contraception during and for 30 days after the study.
* The patient must present with an acute respiratory illness (≤7 days duration) with which history and physical examination is consistent with a diagnosis of CAP.

Patients requiring immediate study drug therapy before serology or culture results are known may be entered with a presumptive diagnosis of CAP based on:

A chest radiograph at baseline, which shows a new infiltrate(s) consistent with pneumonia as interpreted by the radiologist or the investigator and subsequently confirmed by the radiologist.

AND at least 2 of the following signs and symptoms:

New or increased cough. Purulent sputum or change in sputum character. Auscultatory findings consistent with pneumonia. New onset or progressive dyspnea or tachypnea. Fever >38ºC oral or >38.5ºC tympanic. White blood cell (WBC) count greater than 10,000 cells/mm3 or >15% immature neutrophils (bands), regardless of total peripheral WBC count, or less than 4,500 cells/mm3.

Patient must be able to swallow large capsules intact.

A written, voluntarily signed informed consent must be obtained from the patient prior to the initiation of any study-related procedures.

Exclusion Criteria:

* Hypersensitivity to linezolid.
* Patients are excluded if they have taken oral or parenteral antibiotics as follows:

long-acting penicillin within 28 days of enrollment azithromycin, ceftriaxone, or telithromycin within 14 days prior to enrollment any other antibiotics for >24 hours within 3 days of enrollment

* Require parenteral antibiotics for the treatment for CAP.
* Patient should not have been hospitalized or resided in a long-term facility for at least 14 days before the onset of symptoms.
* Evidence of other pulmonary disease that precluded evaluation of therapeutic response. Patients with known bronchial obstruction or a history of postobstructive pneumonia. (This does not exclude patients who have chronic obstructive pulmonary disease).
* Experienced a recent clinically significant coagulopathy.
* History of cystic fibrosis, active tuberculosis, meningitis, endocarditis, or osteomyelitis.
* Immunocompromised patients including, but not limited to patients with a CD4+ cell count of <350 cells/mm3 secondary to human immunodeficiency virus (HIV) infection, neutropenic patients with granulocytes <1000/mm3 or immunosuppression secondary to drugs such as corticosteroid therapy (>10 mg/day of prednisone or equivalent for at least the past 3 months), splenectomized patients or patients with known hyposplenia or asplenia.
* Patients who have severe liver disease.
* Treatment with an investigational drug within 4 weeks prior to study drug administration.
* Any underlying condition or disease state that would interfere with the completion of the study procedures and evaluation of the absorption of study drug.
* Patients with bronchiectasis and a history of recent respiratory infection caused by Pseudomonas aeruginosa.
* Any infection which requires the use of a concomitant antimicrobial agent, in addition to study drug.
* Patients taking serotonergic agents, selective serotonin reuptake inhibitors (SSRIs) or monoamine oxidase inhibitors (MAOIs).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (8):
  - eStudySite, San Diego, California
  - Olive View- UCLA Center, Dept. Emergency Medicine, Sylmar, California
  - Wayne State University School of Medicine/Detroit Receiving Hospital, Detroit, Michigan
  - Arnold Markowitz, MD, Keego Harbor, Michigan
  - Mercury Street Medical Group, LLC, Butte, Montana
  - Dr. John Bernard, Belvidere, New Jersey
  - University of Medicine & Dentistry of New Jersey, School of Osteopathic Medicine (UMDNJ-SOM), Cherry Hill, New Jersey
  - Warminster Medical Associates, P.C., Warminster, Pennsylvania
- Canada (14):
  - Ronald Collette, MD, Burnaby, British Columbia
  - The Medical Arts Health Research Group, Kelowna, British Columbia
  - Westview Research, North Vancouver, British Columbia
  - The Medical Arts Health Research Group, Penticton, British Columbia
  - Maritime Research Center, Bathurst, New Brunswick
  - Source Unique Research, Hawkesbury, Ontario
  - Gordon Schacter, MD, London, Ontario
  - London East Medical Centre, London, Ontario
  - SKDS Research Inc., Newmarket, Ontario
  - University of Ottawa Health Services, Ottawa, Ontario
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Kings County Medical Centre, Montague, Prince Edward Island
  - Rhodin Recherche Clinique, Drummondville, Quebec
  - Centre Medical Acadie, Montreal, Quebec
- Russia (8):
  - Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky, Moscow
  - Moscow State Medico-Stomatological University, Moscow
  - State Healthcare Institution "City Clinical Hospital # 29", Moscow
  - State Healthcare Institution Moscow, Moscow
  - City Hospital # 31, Saint Petersburg
  - St. Petersburg City Hospital # 26, Saint Petersburg
  - St. Petersburg Pavlov State Medical University, Saint Petersburg
  - St. Petersburg Scientific-Research Institute of Pulmonology at State Medical University named after Academician I.P. Pavlov, Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study targeted adult patients with mild to moderate (i.e., CURB-65 score of 0 or 1) community-acquired pneumonia (CAP).
Period: Overall Study
Arm/Group | Radezolid 300 mg PO Daily (QD) | Radezolid 450 mg PO Daily (QD) | Radezolid 450 mg PO Twice Daily (BID)
Started | 53 | 52 | 53
Completed | 45 | 46 | 45
Not Completed | 8 | 6 | 8
Not completed — Adverse Event | 2 | 3 | 2
Not completed — Lack of Efficacy | 0 | 2 | 1
Not completed — Protocol Violation | 2 | 0 | 2
Not completed — Lost to Follow-up | 3 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radezolid 300 mg PO Daily (QD) | Radezolid 450 mg PO Daily (QD) | Radezolid 450 mg PO Twice Daily (BID) | Total
Number analyzed (Participants) | 53 | 52 | 53 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (18.37) | 50.4 (14.55) | 52.1 (15.61) | 50.7 (16.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 22 | 61
  Male | 31 | 35 | 31 | 97
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 17 | 62
  Canada | 14 | 16 | 21 | 51
  Russian Federation | 15 | 15 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure in the Clinically Evaluable (CE) Population at Test of Cure (TOC)
Description: Patients were considered cured if all systemic signs and symptoms of CAP present at screening were improved or resolved and no further antibiotic therapy was necessary. In addition, the follow-up chest X-ray was to be either stable or improved.
Time Frame: Study days 14-38
Population: Clinically evaluable patients were those that had a diagnosis of CAP, as defined in the inclusion criteria; who received an appropriate course of therapy; who did not receive any other concomitant antibiotics, and who returned for a TOC visit in the appropriate time frame.
Measure: Number; unit: Participants
Arm/Group | Radezolid 300 mg PO Daily (QD) | Radezolid 450 mg PO Daily (QD) | Radezolid 450 mg PO Twice Daily (BID)
Number analyzed (Participants) | 37 | 44 | 41
Participants | 34 | 37 | 32

2. Other Pre Specified Outcome: Per Patient Microbiological Response of Eradicated in the Microbiologically Evaluable (ME) Population at Test of Cure (TOC)
Description: The number of ME patients (defined as those CE patients with evidence of 1 or more of 7 key CAP pathogens: S. pneumoniae, H. influenzae, M. catarrhalis, M. pneumoniae, C. pneumoniae, and L. pneumophila) with a microbiologic response of eradicated, i.e. either documented eradication of the baseline pathogen(s), or presumed eradication in the setting of clinical cure with no material to culture.
Time Frame: Study Days 14-38
Population: Microbiologically evaluable (ME) patients were defined as CE patients with evidence of 1 or more of 7 key CAP pathogens: S. pneumoniae, H. influenzae, M. catarrhalis, M. pneumoniae, C. pneumoniae, and L. pneumophila.
Measure: Number; unit: Participants
Arm/Group | Radezolid 300 mg PO Daily (QD) | Radezolid 450 mg PO Daily (QD) | Radezolid 450 mg PO Twice Daily (BID)
Number analyzed (Participants) | 17 | 26 | 26
Participants | 16 | 20 | 18

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were to be reported from the signing of the informed consent until the test of cure (TOC) visit.
Arm/Group | Radezolid 300 mg PO Daily (QD) | Radezolid 450 mg PO Daily (QD) | Radezolid 450 mg PO Twice Daily (BID)
Serious Adverse Events (participants affected / at risk) | 3/53 | 2/52 | 5/53
Other Adverse Events (participants affected / at risk) | 11/53 | 17/52 | 28/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radezolid 300 mg PO Daily (QD) (N=53) | Radezolid 450 mg PO Daily (QD) (N=52) | Radezolid 450 mg PO Twice Daily (BID) (N=53)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dehyrdation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radezolid 300 mg PO Daily (QD) (N=53) | Radezolid 450 mg PO Daily (QD) (N=52) | Radezolid 450 mg PO Twice Daily (BID) (N=53)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 10 (10) | 19 (19)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Fungal infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
The yield of typical bacterial pathogens, most importantly S. pneumoniae, was quite low. The presence of atypical pathogens was assessed only by paired serologies, not by culture or polymerase chain reaction (PCR).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor retains publication rights.